CLINICAL TRIAL: NCT01433627
Title: Phase IIIb Study Minimizing Adverse Haemmhorragic Events by TRansradial Access Site and Systemic Implementation of angioX (MATRIX)
Brief Title: Minimizing Adverse Haemorrhagic Events by TRansradial Access Site and Systemic Implementation of angioX
Acronym: MATRIX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Italian Society of Invasive Cardiology (Other)
Collaborators: Eustrategy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: RFBU 11-I; 2011-000430-11 (EudraCT Number)
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Acute Coronary Syndromes; STEMI; NSTEMI
Keywords: acute coronary syndromes; myocardial infarction; access site; bivalirudin; bleedings
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- trans-radial and short-term Bivalirudin (Experimental): Patients will be randomized to receive a trans-radial intervention and concomitant bivalirudin infusion. bivalirudin will be stopped at the end of PCI.
  Interventions: Other: trans-radial and short-term bivalirudin
- trans-radial and long-term bivalirudin (Experimental): Trans-radial intervention: will be performed according to institutional guidelines and established local practice.
  Bivalirudin: given immediately upon enrolment as bolus of 0.75 mg/kg followed immediately by an infusion of 1.75 mg/kg/h. This infusion should be run continuously until completion of PCI at which time the infusion should be reduced to a dose of 0.25 mg/kg/h for at least 6 hours. An optional higher-dose infusion of 1.75 mg/kg/h is also permitted for up to 4 hours in the prolonged infusion arm but prohibited in the short bivalirudin group.
  Interventions: Other: trans-radial and long-term bivalirudin infusion
- trans-radial and standard of care pharmacology (Experimental): Trans-radial intervention: will be performed according to institutional guidelines and established local practice.
  unfractionated heparin (UFH) which may be followed by the addition of a glycoprotein IIb/IIIa inhibitor
  Interventions: Other: trans-radial and standard of care pharmacology
- trans-femoral and short-term bivalirudin (Experimental): Trans-femoral intervention: will be performed according to institutional guidelines and established local practice. Access closure devices are allowed as per local practice.
  Bivalirudin will be given immediately upon enrolment as bolus of 0.75 mg/kg followed immediately by an infusion of 1.75 mg/kg/h. This infusion should be run continuously until completion of PCI.
  Interventions: Other: Trans-femoral and Short-term bivalirudin
- Trans-femoral and long-term bivalirudin (Experimental): Trans-femoral intervention: will be performed according to institutional guidelines and established local practice. Access closure devices are allowed as per local practice.
  Bivalirudin will be given immediately upon enrolment as bolus of 0.75 mg/kg followed immediately by an infusion of 1.75 mg/kg/h. This infusion should be run continuously until completion of PCI at which time the infusion should be reduced to a dose of 0.25 mg/kg/h for at least 6 hours. An optional higher-dose infusion of 1.75 mg/kg/h is also permitted for up to 4 hours in the prolonged infusion arm but prohibited in the short bivalirudin group.
  Interventions: Other: trans-femoral and long-term bivalirudin infusion
- trans-femoral and standard of care pharmacology (Active Comparator): Trans-femoral intervention: will be performed according to institutional guidelines and established local practice. Access closure devices are allowed as per local practice. Unfractionated heparin (UFH) (100 IU/kg with no glycoprotein IIb/IIIa inhibitor (GPI) and 60 IU/kg with a GPI); +/- routine or bail out eptifibatide (two 180 μg /kg boluses with a 10 minute interval followed by an infusion of 2.0 μg /kg/min for 72-96 hours) or tirofiban (25 μg/kg followed by an infusion of 0.15 μg/kg/min for 18 to 24 hours) or abciximab (bolus of 0.25 mg/kg followed by an infusion of 0.125 μg/kg/min for 12-24 hours (maximum dose, 10 μg/min).
  Interventions: Other: trans-femoral and standard of care pharmacology

INTERVENTIONS:
Other: trans-radial and short-term bivalirudin — trans-radial intervention followed by Bivalirudin given immediately upon enrolment as bolus of 0.75 mg/kg followed immediately by an infusion of 1.75 mg/kg/h. This infusion should be run continuously until completion of PCI at which time the infusion should be stopped.
  Other Names: Access site selection and drug administration
  Arms: trans-radial and short-term Bivalirudin
Other: trans-radial and long-term bivalirudin infusion — Trans-radial intervention: will be performed according to institutional guidelines and established local practice.
  Bivalirudin: given immediately upon enrolment as bolus of 0.75 mg/kg followed immediately by an infusion of 1.75 mg/kg/h. This infusion should be run continuously until completion of PCI at which time the infusion should be reduced to a dose of 0.25 mg/kg/h for at least 6 hours. An optional higher-dose infusion of 1.75 mg/kg/h is also permitted for up to 4 hours in the prolonged infusion arm but prohibited in the short bivalirudin group.
  Other Names: access site selection and drug administration
  Arms: trans-radial and long-term bivalirudin
Other: trans-radial and standard of care pharmacology — Unfractionated heparin (UFH) (100 IU/kg with no glycoprotein IIb/IIIa inhibitor (GPI) and 60 IU/kg with a GPI); +/- routine or bail out eptifibatide (two 180 μg /kg boluses with a 10 minute interval followed by an infusion of 2.0 μg /kg/min for 72-96 hours) or tirofiban (25 μg/kg followed by an infusion of 0.15 μg/kg/min for 18 to 24 hours) or abciximab (bolus of 0.25 mg/kg followed by an infusion of 0.125 μg/kg/min for 12-24 hours (maximum dose, 10 μg/min).
  Other Names: access site and drug administration
  Arms: trans-radial and standard of care pharmacology
Other: Trans-femoral and Short-term bivalirudin — Trans-femoral intervention: will be performed according to institutional guidelines and established local practice. Access closure devices are allowed as per local practice.
  Bivalirudin will be given immediately upon enrolment as bolus of 0.75 mg/kg followed immediately by an infusion of 1.75 mg/kg/h. This infusion should be run continuously until completion of PCI.
  Other Names: access site selection and drug administration
  Arms: trans-femoral and short-term bivalirudin
Other: trans-femoral and long-term bivalirudin infusion — Trans-femoral intervention: will be performed according to institutional guidelines and established local practice. Access closure devices are allowed as per local practice.
  Bivalirudin will be given immediately upon enrolment as bolus of 0.75 mg/kg followed immediately by an infusion of 1.75 mg/kg/h. This infusion should be run continuously until completion of PCI at which time the infusion should be reduced to a dose of 0.25 mg/kg/h for at least 6 hours. An optional higher-dose infusion of 1.75 mg/kg/h is also permitted for up to 4 hours in the prolonged infusion arm but prohibited in the short bivalirudin group.
  Other Names: access site selection and drug administration
  Arms: Trans-femoral and long-term bivalirudin
Other: trans-femoral and standard of care pharmacology — Trans-femoral intervention: will be performed according to institutional guidelines and established local practice. Access closure devices are allowed as per local practice. Unfractionated heparin (UFH) (100 IU/kg with no glycoprotein IIb/IIIa inhibitor (GPI) and 60 IU/kg with a GPI); +/- routine or bail out eptifibatide (two 180 μg /kg boluses with a 10 minute interval followed by an infusion of 2.0 μg /kg/min for 72-96 hours) or tirofiban (25 μg/kg followed by an infusion of 0.15 μg/kg/min for 18 to 24 hours) or abciximab (bolus of 0.25 mg/kg followed by an infusion of 0.125 μg/kg/min for 12-24 hours (maximum dose, 10 μg/min).
  Other Names: access site selection and drug administration
  Arms: trans-femoral and standard of care pharmacology

SUMMARY:
This protocol describes a study to compare intended trans-radial versus trans-femoral intervention and bivalirudin monotherapy versus current European standard of care consisting of unfractionated heparin (UFH) plus provisional use of glycoprotein IIb/IIIa inhibition via the use of one of the three available agents on the market (e.g. abciximab, tirofiban or eptifibatide) in patients (≥18 years) with ACS, that are intended for an invasive management strategy. This study will be conducted in compliance with Good Clinical Practices (GCP) including the Declaration of Helsinki and all applicable regulatory requirements.

DETAILED DESCRIPTION:
The use of combined antithrombotic therapies over the last two decades has decreased the risk of a heart attack after percutaneous coronary intervention substantially but has also been associated with a significant increase in bleeding risk. Therapies or strategies that maintain the benefits seen with currently available antithrombotic therapies but which have lower bleeding risk are therefore of great clinical importance. Indeed, major bleeding is currently the most common non-cardiac complication of therapy for patients with coronary artery disease who have undergone percutaneous coronary intervention (PCI).

Bleeding in patients with acute coronary syndrome (ACS) is associated with an increased risk of long term mortality and morbidity, and this relationship is currently thought to be causal. Therefore' reducing the frequency of bleeding events while maintaining efficacy is an important goal in the management of patients with ACS. The most common site of bleeding in invasively managed patients with ACS is at the femoral artery puncture site used for heart catheterization

The MATRIX study is a multi-centre, prospective, randomised, open-label, 2 by 2 factorial comparison of trans-radial vs. trans-femoral intervention and bivalirudin vs. unfractionated heparin and provisional use of glycoprotein IIb/IIIa inhibitor.

Objectives:

1. To demonstrate that trans-radial intervention as compared to femoral access site is associated to lower rate of the composite endpoint of death, MI or stroke within the first 30 days after randomization in acute coronary syndrome patients undergoing early invasive management.
2. To demonstrate that bivalirudin infusion as compared to standard of care therapy consisting of unfractionated heparin and provisional use of glycoprotein IIb/IIIa inhibitors are associated to lower rate of the composite endpoint of death, MI or stroke within the first 30 days after randomization in acute coronary syndrome patients undergoing early invasive management.

Patients randomly assigned to receive bivalirudin will be randomized to stop bivalirudin infusion at the end of PCI or to prolong bivalirudin at an infusion rate of 0.25 mg/kg/hour for at least 6 hours after completion of PCI. The primary hypothesis in this sub-randomization is that prolonged post-intervention bivalirudin infusion will be superior to no bivalirudin post-PCI infusion with respect to the net composite outcome consisting of any death, MI, stroke, urgent TVR, stent thrombosis and BARC-defined type 3 and 5 bleeding events within 30 days. Secondary objectives for the sub-randomization of prolonged bivalirudin versus no post-PCI infusion in the bivalirudin group will consist of each component of the primary composite endpoint through the entire follow-up duration

ELIGIBILITY:
Inclusion Criteria:

NSTEACS definition: Patients with all of the following criteria will be eligible:

1. history consistent with new, or worsening ischemia, occurring at rest or with minimal activity;
2. enrollment within 7 days of the most recent symptoms;
3. planned coronary angiography with possible indication to PCI;
4. at least 2 of the following criteria: 1. Aged 60 years or older, 2. Troponin T or I or creatine kinase MB above the upper limit of normal; 3. Electrocardiograph changes compatible with ischemia, ie, ST depression of 1 mm or greater in 2 contiguous leads, T-wave inversion more than 3 mm, or any dynamic ST shifts;

STEMI definition: i) chest pain for >20 min with an electrocardiographic ST-segment elevation ≥1 mm in two or more contiguous electrocardiogram (ECG) leads, or with a new left bundle-branch block, or an infero-lateral myocardial infarction (MI) with ST segment depression of ≥1 mm in ≥2 of leads V1-3 with a positive terminal T wave and ii) admission either within 12 h of symptom onset or between 12 and 24 h after onset with evidence of continuing ischemia or previous lytic treatment.

Exclusion Criteria:

1. Patients who can not give informed consent or have a life expectancy of <30 days
2. Allergy/intolerance to Bivalirudin or unfractionated heparin.
3. Stable or silent CAD as indication to coronary angiography
4. Treatment with LWMH within the past 6 hours
5. Treatment with any GPI in the previous 3 days
6. Absolute contraindications or allergy that cannot be pre-medicated to iodinated contrast or to any of the study medications including aspirin or clopidogrel.
7. Contraindications to angiography, including but not limited to severe peripheral vascular disease.
8. If it is known pregnant or nursing mothers. Women of child-bearing age will be asked if they are pregnant or think that they may be pregnant.
9. If it is known a creatinine clearance <30 mL/min or dialysis dependent.
10. Previous enrollment in this study.
11. Treatment with other investigational drugs or devices within the 30 days preceding
12. Randomisation or planned use of other investigational drugs or devices in this trial.
13. Severe uncontrolled hypertension (defined as persistent systolic blood pressure higher than 220 mmHg despite medical treatment).
14. Subacute bacterial endocarditis
15. PCI in the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7200 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
the composite of Death, non-fatal myocardial infarction or stroke | 30 days
  To demonstrate in ACS patients undergoing an early invasive management, i.e. diagnostic coronary angiogram+PCI or ad hoc planned PCI that trans-radial intervention as compared to femoral access site is associated to lower rate of the composite endpoint of death, MI or stroke within the first 30 days after randomization.
The composite of death, non-fatal myocardial infarction or stroke | 30 days
  To demonstrate that in an ACS patients with an intended PCI treatment strategy or in whom upstream treatment was felt necessary by local investigators the use of bivalirudin as compared to unfractionated heparin (UFH) plus or minus Glycoprotein IIb/IIIa inhibitor (GPI) is associated to lower rate of the composite endpoint of death, MI or stroke within the first 30 days after randomization.
Death, non-fatal myocardial infarction, stroke, stent thrombosis or BARC-defined type 3 or 5 bleedings | 30 days
  The primary hypothesis of this sub-randomization is that prolonged post-intervention bivalirudin infusion (long bivalirudin arm) will be superior to peri-PCI bivalirudin infusion only (short bivalirudin arm) with respect to the net composite outcomes consisting of any death, MI, stroke, stent thrombosis or BARC-defined type 3 and 5 bleeding events within 30 days.

SECONDARY OUTCOMES:
the composite endpoint of death, MI, stroke or BARC-defined type 3 and 5 major bleeding complications | 30 days
  Key secondary objective: To demonstrate that trans-radial intervention as compared to femoral access site is associated to lower rate of the composite endpoint of death, MI, stroke or BARC-defined type 3 and 5 major bleeding complications within the first 30 days after randomization.
Death, non-fatal MI, stroke or BARC-defined type 3 and 5 major bleeding | 30 days
  To demonstrate that use of bivalirudin as compared to unfractionated heparin (UFH) plus or minus Glycoprotein IIb/IIIa inhibitor (GPI) is associated to lower rate of the composite endpoint of death, MI, stroke or BARC-defined type 3 and 5 major bleeding complications within the first 30 days after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Valgimigli, MD PhD, Principal Investigator — Erasmus MC, Thoraxcenter, The Netherlands
Locations (62):
- Italy (62):
  - Ospedale Clinicizzato SS Annunziata di Chieti, Chieti, Abruzzo
  - Ospedale Civile Santo Spirito, Pescara, Abruzzo
  - Ospedale Di Venere - ASL Bari, Bari, Apulia
  - Città di Lecce Ospedale (GVM), Lecce, Apulia
  - Ospedale Vito Fazzi, Lecce, Apulia
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Apulia
  - Casa di Cura Villa Verde, Taranto, Apulia
  - Azienda Ospedaliera Pugliese Ciaccio - Catanzaro, Catanzaro, Calabria
  - A.O. AORN Cardarelli, Napoli, Campania
  - Azienda Ospedaliera Monaldi, Napoli, Campania
  - Policlinico Federico II, Napoli, Campania
  - Policlinico Sant'Orsola Malpighi, Bologna, Emilia-Romagna
  - University Hospital of Ferrara, Ferrara, Emilia-Romagna
  - Ospedale G. B. Morgagni, Forlì, Emilia-Romagna
  - Azienda S. Maria Nuova di Reggio Emilia, Reggio Emilia, Emilia-Romagna
  - Ospedale degli Infermi, Rimini, Emilia-Romagna
  - Azienda Ospedaliera Universitaria Ospedali Riuniti, Trieste, Friuli Venezia Giulia
  - Azienda Ospedaliera S. Maria della Misericordia di Udine, Udine, Friuli Venezia Giulia
  - Ospedale Santa Maria Goretti, Latina, Lazio
  - A.O. Sandro Pertini, Rome, Lazio
  - Ospedale del Santo Spirito in Sassia, Rome, Lazio
  - Ospedale San Camillo di Roma, Rome, Lazio
  - Policlinico Casilino, Rome, Lazio
  - Azienda Ospedaliera Universitaria "San Martino", Genoa, Liguria
  - Ospedale Villa Scassi, Genoa, Liguria
  - Spedali Civili di Brescia, Brescia, Lombardy
  - Azienda Ospedaliera Sant'Anna di Como, Como, Lombardy
  - Azienda Ospedaliera di Desio e Vimercate - P.O. di Desio, Desio, Lombardy
  - Ospedale Sacra Famiglia, Erba, Lombardy
  - Ospedale di Lodi, Lodi, Lombardy
  - A.O: Fatebenefratelli e oftalmico, Milan, Lombardy
  - IRCCS Multimedica, Sesto San Giovanni, Lombardy
  - A.O. Treviglio, Treviglio, Lombardy
  - A. O. Ospedale Civile di Vimercate, Vimercate, Lombardy
  - Policlinico San Marco, Zingonia, Lombardy
  - Istituto Clinico Humanitas IRCCS, Rozzano, MI
  - Ospedale S. Croce e Carlo, Cuneo, Piedmont
  - Azienda Ospedaliero-Universitaria "Maggiore della Carità", Novara, Piedmont
  - A. O. Universitaria San Luigi Gonzaga di Orbassano, Orbassano, Piedmont
  - Ospedali Riuniti ASL 17, Savigliano, Piedmont
  - A.O. Universitaria Molinette San Giovanni Battista, Turin, Piedmont
  - Ospedale San Giovanni Bosco, Turin, Piedmont
  - Maria Cecilia Hospital, Cotignola, RA
  - Azienda USL Sirai, Carbonia, Sardinia
  - Ospedale San Francesco, Nuoro, Sardinia
  - A. O. Universitaria Policlinico V. Emanuele Ferrarotto, Catania, Sicily
  - Villa Maria Eleonora Hospital, Palermo, Sicily
  - A.O. Civili Riuniti - Giovanni Paolo II, Sciacca, Sicily
  - Ospedale Umberto I di Siracusa, Syracuse, Sicily
  - Ospedale S. Vincenzo, Taormina, Sicily
  - A.O. G. Mazzoni, Ascoli Piceno, The Marches
  - Azienda Ospedaliera San Salvatore, Pesaro, The Marches
  - Ospedale degli Infermi, Rivoli, TO
  - Presidio Ospedaliero Santa Chiara, Trento, Trentino-Alto Adige
  - P.O. Zona Aretina-Ospedale San Donato, Arezzo, Tuscany
  - Azienda USL - Grosseto, Grosseto, Tuscany
  - Ospedale del Cuore "G. Pasquinucci" Massa, Massa Carrara, Tuscany
  - Azienda Ospedaliera Universitaria Pisana, Pisa, Tuscany
  - Presidio Ospedaliero di Este, Este, Veneto
  - Ospedale Mater Salutis di Legnago, Legnago, Veneto
  - Ospedale Civile di Mirano, Mirano, Veneto
  - Università Campus Bio-Medico di Roma, Rome

REFERENCES:
- [Derived] Leonardi S, Landi A, Zito A, Branca M, Frigoli E, Ando' G, Briguori C, Calabro P, Gagnor A, Garbo R, Heg D, Limbruno U, Milzi A, Omerovic E, Russo F, Sabate M, Santarelli A, Sardella G, Tosi P, Van't Hof AWJ, Vranckx P, Valgimigli M. Prognostic Implications of Evolving Universal Definitions of Periprocedural Myocardial Infarction in Patients With Acute Coronary Syndrome. Circulation. 2026 Jan 27;153(4):230-242. doi: 10.1161/CIRCULATIONAHA.125.077174. Epub 2026 Jan 6. PMID 41493005
- [Derived] Landi A, Zito A, Singh M, Angiolillo DJ, Capodanno D, Frigoli E, Milzi A, Rao SV, Urban P, Valgimigli M. Validation of the Mayo Clinic Percutaneous Coronary Intervention Risk Prediction Score in Patients With Acute Coronary Syndrome. J Am Heart Assoc. 2025 Oct 21;14(20):e043012. doi: 10.1161/JAHA.125.043012. Epub 2025 Oct 9. PMID 41065238
- [Derived] Landi A, Chiarito M, Branca M, Frigoli E, Gagnor A, Calabro P, Briguori C, Ando G, Repetto A, Limbruno U, Sganzerla P, Lupi A, Cortese B, Ausiello A, Ierna S, Esposito G, Ferrante G, Santarelli A, Sardella G, Varbella F, Heg D, Mehran R, Valgimigli M. Validation of a Contemporary Acute Kidney Injury Risk Score in Patients With Acute Coronary Syndrome. JACC Cardiovasc Interv. 2023 Aug 14;16(15):1873-1886. doi: 10.1016/j.jcin.2023.06.015. PMID 37587595
- [Derived] Garg M, Garcia-Garcia HM, Calderon AT, Gupta J, Sortur S, Levine MB, Singla P, Picchi A, Sardella G, Adamo M, Frigoli E, Limbruno U, Rigattieri S, Diletti R, Boccuzzi G, Zimarino M, Contarini M, Russo F, Calabro P, Ando G, Varbella F, Garducci S, Palmieri C, Briguori C, Sanchez JS, Valgimigli M. Reproducibility of an artificial intelligence optical coherence tomography software for tissue characterization: Implications for the design of longitudinal studies. Cardiovasc Revasc Med. 2024 Jan;58:79-87. doi: 10.1016/j.carrev.2023.07.003. Epub 2023 Jul 16. PMID 37474355
- [Derived] Landi A, Branca M, Leonardi S, Frigoli E, Vranckx P, Tebaldi M, Varbella F, Calabro P, Esposito G, Sardella G, Garducci S, Ando G, Limbruno U, Sganzerla P, Santarelli A, Briguori C, Colangelo S, Brugaletta S, Adamo M, Omerovic E, Heg D, Windecker S, Valgimigli M; MATRIX Investigators. Transient vs In-Hospital Persistent Acute Kidney Injury in Patients With Acute Coronary Syndrome. JACC Cardiovasc Interv. 2023 Jan 23;16(2):193-205. doi: 10.1016/j.jcin.2022.10.009. Epub 2022 Dec 28. PMID 36697156
- [Derived] Dan K, Garcia-Garcia HM, Yacob O, Kuku KO, Diaz-Torres MA, Picchi A, Sardella G, Adamo M, Frigoli E, Limbruno U, Rigattieri S, Diletti R, Boccuzzi G, Zimarino M, Contarini M, Russo F, Calabro P, Ando G, Varbella F, Garducci S, Palmieri C, Briguori C, Karagiannis A, Dijkstra J, Valgimigli M. Ultra-Short Term Evaluation of Coronary Vessel Wall Changes in Reference Segments Adjacent to Culprit Lesions in ST-Segment Elevation Myocardial Infarction. J Invasive Cardiol. 2021 Dec;33(12):E923-E930. doi: 10.25270/jic/21.00035. Epub 2021 Nov 18. PMID 34792483
- [Derived] Landi A, Branca M, Ando G, Russo F, Frigoli E, Gargiulo G, Briguori C, Vranckx P, Leonardi S, Gragnano F, Calabro P, Campo G, Ambrosio G, Santucci A, Varbella F, Zaro T, Heg D, Windecker S, Juni P, Pedrazzini G, Valgimigli M; MATRIX Investigators. Acute kidney injury in patients with acute coronary syndrome undergoing invasive management treated with bivalirudin vs. unfractionated heparin: insights from the MATRIX trial. Eur Heart J Acute Cardiovasc Care. 2021 Dec 18;10(10):1170-1179. doi: 10.1093/ehjacc/zuab080. PMID 34491323
- [Derived] Gragnano F, Branca M, Frigoli E, Leonardi S, Vranckx P, Di Maio D, Monda E, Fimiani L, Fioretti V, Chianese S, Esposito F, Franzese M, Scalise M, D'Angelo C, Scalise R, De Blasi G, Ando G, Esposito G, Calabro P, Windecker S, Pedrazzini G, Valgimigli M; MATRIX Trial Investigators. Access-Site Crossover in Patients With Acute Coronary Syndrome Undergoing Invasive Management. JACC Cardiovasc Interv. 2021 Feb 22;14(4):361-373. doi: 10.1016/j.jcin.2020.11.042. PMID 33602431
- [Derived] Leonardi S, Gragnano F, Carrara G, Gargiulo G, Frigoli E, Vranckx P, Di Maio D, Spedicato V, Monda E, Fimiani L, Fioretti V, Esposito F, Avvedimento M, Magliulo F, Leone A, Chianese S, Franzese M, Scalise M, Schiavo A, Mazzone P, Esposito G, Ando G, Calabro P, Windecker S, Valgimigli M. Prognostic Implications of Declining Hemoglobin Content in Patients Hospitalized With Acute Coronary Syndromes. J Am Coll Cardiol. 2021 Feb 2;77(4):375-388. doi: 10.1016/j.jacc.2020.11.046. PMID 33509394
- [Derived] Gargiulo G, Valgimigli M, Sunnaker M, Vranckx P, Frigoli E, Leonardi S, Spirito A, Gragnano F, Manavifar N, Galea R, De Caterina AR, Calabro P, Esposito G, Windecker S, Hunziker L. Choice of access site and type of anticoagulant in acute coronary syndromes with advanced Killip class or out-of-hospital cardiac arrest. Rev Esp Cardiol (Engl Ed). 2020 Nov;73(11):893-901. doi: 10.1016/j.rec.2020.01.005. Epub 2020 Mar 6. English, Spanish. PMID 32151464
- [Derived] Garcia-Garcia HM, Picchi A, Sardella G, Adamo M, Frigoli E, Limbruno U, Rigattieri S, Diletti R, Boccuzzi G, Zimarino M, Contarini M, Russo F, Calabro' P, Ando G, Varbella F, Garducci S, Palmieri C, Briguori C, Kuku KO, Rothenbuhler M, Karagiannis A, Valgimigli M. Comparison of intra-procedural vs. post-stenting prolonged bivalirudin infusion for residual thrombus burden in patients with ST-segment elevation myocardial infarction undergoing: the MATRIX (Minimizing Adverse Haemorrhagic Events by TRansradial Access Site and angioX) OCT study. Eur Heart J Cardiovasc Imaging. 2019 Dec 1;20(12):1418-1428. doi: 10.1093/ehjci/jez040. PMID 30920584
- [Derived] Gargiulo G, Carrara G, Frigoli E, Leonardi S, Vranckx P, Campo G, Varbella F, Calabro P, Zaro T, Bartolini D, Briguori C, Ando G, Ferrario M, Limbruno U, Colangelo S, Sganzerla P, Russo F, Nazzaro MS, Esposito G, Ferrante G, Santarelli A, Sardella G, Windecker S, Valgimigli M. Post-Procedural Bivalirudin Infusion at Full or Low Regimen in Patients With Acute Coronary Syndrome. J Am Coll Cardiol. 2019 Feb 26;73(7):758-774. doi: 10.1016/j.jacc.2018.12.023. PMID 30784669
- [Derived] Valgimigli M, Frigoli E, Leonardi S, Vranckx P, Rothenbuhler M, Tebaldi M, Varbella F, Calabro P, Garducci S, Rubartelli P, Briguori C, Ando G, Ferrario M, Limbruno U, Garbo R, Sganzerla P, Russo F, Nazzaro M, Lupi A, Cortese B, Ausiello A, Ierna S, Esposito G, Ferrante G, Santarelli A, Sardella G, de Cesare N, Tosi P, van 't Hof A, Omerovic E, Brugaletta S, Windecker S, Heg D, Juni P; MATRIX Investigators. Radial versus femoral access and bivalirudin versus unfractionated heparin in invasively managed patients with acute coronary syndrome (MATRIX): final 1-year results of a multicentre, randomised controlled trial. Lancet. 2018 Sep 8;392(10150):835-848. doi: 10.1016/S0140-6736(18)31714-8. Epub 2018 Aug 25. PMID 30153988
- [Derived] Gargiulo G, Carrara G, Frigoli E, Vranckx P, Leonardi S, Ciociano N, Campo G, Varbella F, Calabro P, Garducci S, Iannone A, Briguori C, Ando G, Crimi G, Limbruno U, Garbo R, Sganzerla P, Russo F, Lupi A, Cortese B, Ausiello A, Ierna S, Esposito G, Zavalloni D, Santarelli A, Sardella G, Tresoldi S, de Cesare N, Sciahbasi A, Zingarelli A, Tosi P, van 't Hof A, Omerovic E, Brugaletta S, Windecker S, Valgimigli M. Bivalirudin or Heparin in Patients Undergoing Invasive Management of Acute Coronary Syndromes. J Am Coll Cardiol. 2018 Mar 20;71(11):1231-1242. doi: 10.1016/j.jacc.2018.01.033. PMID 29544607
- [Derived] Gargiulo G, Ariotti S, Vranckx P, Leonardi S, Frigoli E, Ciociano N, Tumscitz C, Tomassini F, Calabro P, Garducci S, Crimi G, Ando G, Ferrario M, Limbruno U, Cortese B, Sganzerla P, Lupi A, Russo F, Garbo R, Ausiello A, Zavalloni D, Sardella G, Esposito G, Santarelli A, Tresoldi S, Nazzaro MS, Zingarelli A, Petronio AS, Windecker S, da Costa BR, Valgimigli M. Impact of Sex on Comparative Outcomes of Radial Versus Femoral Access in Patients With Acute Coronary Syndromes Undergoing Invasive Management: Data From the Randomized MATRIX-Access Trial. JACC Cardiovasc Interv. 2018 Jan 8;11(1):36-50. doi: 10.1016/j.jcin.2017.09.014. PMID 29301646
- [Derived] Ando G, Cortese B, Russo F, Rothenbuhler M, Frigoli E, Gargiulo G, Briguori C, Vranckx P, Leonardi S, Guiducci V, Belloni F, Ferrari F, de la Torre Hernandez JM, Curello S, Liistro F, Perkan A, De Servi S, Casu G, Dellavalle A, Fischetti D, Micari A, Loi B, Mangiacapra F, Russo N, Tarantino F, Saia F, Heg D, Windecker S, Juni P, Valgimigli M; MATRIX Investigators. Acute Kidney Injury After Radial or Femoral Access for Invasive Acute Coronary Syndrome Management: AKI-MATRIX. J Am Coll Cardiol. 2017 May 11:S0735-1097(17)36897-3. doi: 10.1016/j.jacc.2017.02.070. Online ahead of print. PMID 28528767
- [Derived] Leonardi S, Frigoli E, Rothenbuhler M, Navarese E, Calabro P, Bellotti P, Briguori C, Ferlini M, Cortese B, Lupi A, Lerna S, Zavallonito-Parenti D, Esposito G, Tresoldi S, Zingarelli A, Rigattieri S, Palmieri C, Liso A, Abate F, Zimarino M, Comeglio M, Gabrielli G, Chieffo A, Brugaletta S, Mauro C, Van Mieghem NM, Heg D, Juni P, Windecker S, Valgimigli M; MATRIX Investigators. Bivalirudin or unfractionated heparin in patients with acute coronary syndromes managed invasively with and without ST elevation (MATRIX): randomised controlled trial. BMJ. 2016 Sep 27;354:i4935. doi: 10.1136/bmj.i4935. PMID 27677503
- [Derived] Valgimigli M, Frigoli E, Leonardi S, Rothenbuhler M, Gagnor A, Calabro P, Garducci S, Rubartelli P, Briguori C, Ando G, Repetto A, Limbruno U, Garbo R, Sganzerla P, Russo F, Lupi A, Cortese B, Ausiello A, Ierna S, Esposito G, Presbitero P, Santarelli A, Sardella G, Varbella F, Tresoldi S, de Cesare N, Rigattieri S, Zingarelli A, Tosi P, van 't Hof A, Boccuzzi G, Omerovic E, Sabate M, Heg D, Juni P, Vranckx P; MATRIX Investigators. Bivalirudin or Unfractionated Heparin in Acute Coronary Syndromes. N Engl J Med. 2015 Sep 10;373(11):997-1009. doi: 10.1056/NEJMoa1507854. Epub 2015 Sep 1. PMID 26324049
- [Derived] Ando G, Cortese B, Frigoli E, Gagnor A, Garducci S, Briguori C, Rubartelli P, Calabro P, Valgimigli M; MATRIX investigators. Acute kidney injury after percutaneous coronary intervention: Rationale of the AKI-MATRIX (acute kidney injury-minimizing adverse hemorrhagic events by TRansradial access site and systemic implementation of angioX) sub-study. Catheter Cardiovasc Interv. 2015 Nov;86(5):950-7. doi: 10.1002/ccd.25932. Epub 2015 Apr 9. PMID 25854692
- [Derived] Valgimigli M, Gagnor A, Calabro P, Frigoli E, Leonardi S, Zaro T, Rubartelli P, Briguori C, Ando G, Repetto A, Limbruno U, Cortese B, Sganzerla P, Lupi A, Galli M, Colangelo S, Ierna S, Ausiello A, Presbitero P, Sardella G, Varbella F, Esposito G, Santarelli A, Tresoldi S, Nazzaro M, Zingarelli A, de Cesare N, Rigattieri S, Tosi P, Palmieri C, Brugaletta S, Rao SV, Heg D, Rothenbuhler M, Vranckx P, Juni P; MATRIX Investigators. Radial versus femoral access in patients with acute coronary syndromes undergoing invasive management: a randomised multicentre trial. Lancet. 2015 Jun 20;385(9986):2465-76. doi: 10.1016/S0140-6736(15)60292-6. Epub 2015 Mar 16. PMID 25791214
- [Derived] Valgimigli M; MATRIX investigators. Design and rationale for the Minimizing Adverse haemorrhagic events by TRansradial access site and systemic Implementation of angioX program. Am Heart J. 2014 Dec;168(6):838-45.e6. doi: 10.1016/j.ahj.2014.08.013. Epub 2014 Sep 16. PMID 25458646
- [Derived] Sciahbasi A, Calabro P, Sarandrea A, Rigattieri S, Tomassini F, Sardella G, Zavalloni D, Cortese B, Limbruno U, Tebaldi M, Gagnor A, Rubartelli P, Zingarelli A, Valgimigli M. Randomized comparison of operator radiation exposure comparing transradial and transfemoral approach for percutaneous coronary procedures: rationale and design of the minimizing adverse haemorrhagic events by TRansradial access site and systemic implementation of angioX - RAdiation Dose study (RAD-MATRIX). Cardiovasc Revasc Med. 2014 Jun;15(4):209-13. doi: 10.1016/j.carrev.2014.03.010. Epub 2014 Mar 26. PMID 24746599
- [Derived] Valgimigli M, Calabro P, Cortese B, Frigoli E, Garducci S, Rubartelli P, Ando G, Santarelli A, Galli M, Garbo R, Repetto A, Ierna S, Briguori C, Limbruno U, Violini R, Gagnor A; MATRIX investigators. Scientific foundation and possible implications for practice of the Minimizing Adverse Haemorrhagic Events by Transradial Access Site andSystemic Implementation of AngioX (MATRIX) trial. J Cardiovasc Transl Res. 2014 Feb;7(1):101-11. doi: 10.1007/s12265-013-9537-1. Epub 2014 Jan 7. PMID 24395497